CLINICAL TRIAL: NCT03051620
Title: Predictive Value of Bone Turnover Markers During Discontinuation With Alendronate
Acronym: PROSA
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Anne Sophie Sølling, MD, PhD student, Aarhus University Hospital
Other Study IDs: 2016-003110-27
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Osteoporosis
Keywords: Bone turnover markers; Alendronate; Drug Holiday
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Discontinue alendronate — 136 patients with osteoporosis stopping treatment with alendronate.

SUMMARY:
The study is a cohort study comprising 136 patients with osteoporosis stopping treatment with alendronate. The study will contribute with new knowledge about biochemical markers of bone turnover as predictors of bone loss after stopping treatment with alendronate.

DETAILED DESCRIPTION:
Background:

Osteoporosis increases the risk of fractures. Alendronate reduces the risk of both vertebral- and hip fractures by approximately 50%. It has, however, become evident that long-term anti-resorptive may lead to serious side effects such as atypical femoral fractures or osteonecrosis of the jaw. The alendronate extension study (FLEX) showed that despite stopping treatment after five years the anti-fracture efficacy regarding non-vertebral and radiological vertebral fractures persists for an additional five years in patients with bone mineral density (BMD) T-score > -2.5 at the femoral neck, no fractures during treatment, and no previous vertebral fracture. It is therefore now clinical practice, that treatment is discontinued after five years in patients that fulfil these criteria. Based on the alendronate extension study it was assumed, that bone turnover monitored by biochemical markers would stay suppressed for years after stopping treatment, however, other studies have demonstrated that there is a great variability in the change in bone turnover markers seen after stopping treatment with alendronate in a real-life setting.

Aim:

To investigate the predictive value of markers of bone turnover on bone loss 12 months after stopping alendronate therapy.

Methods:

The study is a cohort study comprising 136 patients with osteoporosis stopping treatment with alendronate.

Perspectives:

The study will contribute with new knowledge about biochemical markers of bone turnover as predictors of bone loss after stopping treatment with alendronate. It will thus be possible to identify patients who will experience a decrease in BMD during treatment break, and for this particular group of patients treatment can be re-initiated earlier so further loss of bone will be avoided. On the other hand, the biochemical markers of bone turnover could also shed light on who can tolerate treatment break, thereby avoid long-term treatment with alendronate, which may be associated with serious side effects. Finally, the use of blood samples rather than DXA will reduce the use of X-rays.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (postmenopausal for at least two years)
* Men above 50 years
* Treatment for at least five years with alendronate
* BMD T-score total hip > -2.5
* BMD T-score lumbar spine (L1-L4) > -4

Exclusion Criteria:

* Any low-energy fracture within the previous five years during alendronate treatment (not including fingers, toes, or skull)
* Low-energy vertebral fracture at any time
* Low-energy hip fracture at any time
* Ongoing treatment with glucocorticoids
* Metabolic bone disease
* Hormone replacement therapy
* Cancer
* Other conditions affecting bone metabolism

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 140 patients with osteoporosis stopping treatment with alendronate.
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bente L Langdahl, MD PhD DMSc, Study Director — Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Denmark
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Black DM, Cummings SR, Karpf DB, Cauley JA, Thompson DE, Nevitt MC, Bauer DC, Genant HK, Haskell WL, Marcus R, Ott SM, Torner JC, Quandt SA, Reiss TF, Ensrud KE. Randomised trial of effect of alendronate on risk of fracture in women with existing vertebral fractures. Fracture Intervention Trial Research Group. Lancet. 1996 Dec 7;348(9041):1535-41. doi: 10.1016/s0140-6736(96)07088-2. PMID 8950879
- [Background] Liberman UA, Weiss SR, Broll J, Minne HW, Quan H, Bell NH, Rodriguez-Portales J, Downs RW Jr, Dequeker J, Favus M. Effect of oral alendronate on bone mineral density and the incidence of fractures in postmenopausal osteoporosis. The Alendronate Phase III Osteoporosis Treatment Study Group. N Engl J Med. 1995 Nov 30;333(22):1437-43. doi: 10.1056/NEJM199511303332201. PMID 7477143
- [Background] Shane E, Burr D, Ebeling PR, Abrahamsen B, Adler RA, Brown TD, Cheung AM, Cosman F, Curtis JR, Dell R, Dempster D, Einhorn TA, Genant HK, Geusens P, Klaushofer K, Koval K, Lane JM, McKiernan F, McKinney R, Ng A, Nieves J, O'Keefe R, Papapoulos S, Sen HT, van der Meulen MC, Weinstein RS, Whyte M; American Society for Bone and Mineral Research. Atypical subtrochanteric and diaphyseal femoral fractures: report of a task force of the American Society for Bone and Mineral Research. J Bone Miner Res. 2010 Nov;25(11):2267-94. doi: 10.1002/jbmr.253. PMID 20842676
- [Background] Khosla S, Burr D, Cauley J, Dempster DW, Ebeling PR, Felsenberg D, Gagel RF, Gilsanz V, Guise T, Koka S, McCauley LK, McGowan J, McKee MD, Mohla S, Pendrys DG, Raisz LG, Ruggiero SL, Shafer DM, Shum L, Silverman SL, Van Poznak CH, Watts N, Woo SB, Shane E; American Society for Bone and Mineral Research. Bisphosphonate-associated osteonecrosis of the jaw: report of a task force of the American Society for Bone and Mineral Research. J Bone Miner Res. 2007 Oct;22(10):1479-91. doi: 10.1359/jbmr.0707onj. PMID 17663640
- [Background] Black DM, Schwartz AV, Ensrud KE, Cauley JA, Levis S, Quandt SA, Satterfield S, Wallace RB, Bauer DC, Palermo L, Wehren LE, Lombardi A, Santora AC, Cummings SR; FLEX Research Group. Effects of continuing or stopping alendronate after 5 years of treatment: the Fracture Intervention Trial Long-term Extension (FLEX): a randomized trial. JAMA. 2006 Dec 27;296(24):2927-38. doi: 10.1001/jama.296.24.2927. PMID 17190893
- [Background] Schwartz AV, Bauer DC, Cummings SR, Cauley JA, Ensrud KE, Palermo L, Wallace RB, Hochberg MC, Feldstein AC, Lombardi A, Black DM; FLEX Research Group. Efficacy of continued alendronate for fractures in women with and without prevalent vertebral fracture: the FLEX trial. J Bone Miner Res. 2010 May;25(5):976-82. doi: 10.1002/jbmr.11. PMID 20200926
- [Derived] Solling AS, Harslof T, Bruun NH, Langdahl B. The predictive value of bone turnover markers during discontinuation of alendronate: the PROSA study. Osteoporos Int. 2021 Aug;32(8):1557-1566. doi: 10.1007/s00198-021-05835-4. Epub 2021 Jan 30. PMID 33517477

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Population: Postmenopausal women (postmenopausal for at least 2 years) and men above 50 years, who had been treated with alendronate for at least five years and had a total hip bone mineral density (BMD) T-score > -2.5 and lumbar spine BMD (L1-L4) T-score > -4.
  We excluded patients with any low-energy fracture within the previous 5 years during alendronate treatment (not including fingers, toes, or skull), low-energy vertebral fracture or hip fracture at any time, on-going treatment with systemic glucocorticoids, metabolic bone disease, hormone replacement therapy, cancer and other conditions affecting bone metabolism.
Period: Overall Study
Arm/Group | Study Population
Started | 142
Completed | 124
Not Completed | 18
Not completed — Lost to Follow-up | 6
Not completed — n=124 enrolled in extension (all completed) | 12

BASELINE CHARACTERISTICS:
Groups:
- Study Population: Postmenopausal women and men
Arm/Group | Study Population
Number analyzed (Participants) | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 142
  Unknown or Not Reported | 0
Bone mineral density (BMD) lumbar spine [Mean (Standard Deviation); unit: g/cm3] | 0.806 (0.09)
Bone mineral density (BMD) total hip [Mean (Standard Deviation); unit: g/cm3] | 0.780 (0.09)
Baseline CTX [Mean (Standard Deviation); unit: ug/L] | 0.21 (0.1)
Baseline PINP [Mean (Standard Deviation); unit: ug/L] | 28 (9.5)

OUTCOME MEASURES:

1. Primary Outcome: If Carboxy-terminal Collagen Crosslinks (CTX) Three and Six Months After Stopping Alendronate Predicted TH BMD (Total Hip BMD) Loss Above the Least Significant Change at Month 12 at the Individual Level.
Description: We constructed receiver operating characteristic (ROC) curves to evaluate if carboxy-terminal collagen crosslinks (CTX) three and six months after stopping alendronate predicted TH BMD loss above the least significant change (LSC) at month 12 at the individual level.
Time Frame: Baseline and one year after baseline
Population: None of the ROC curves investigating the ability of change in CTX to predict BMD loss beyond LSC at any site at month 12 at the individual level had AUC above 60% meaning that it was not possible to identify a specific cut-off value that could predict significant bone loss at the individual level.
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Study Population: Study population
Arm/Group | Study Population
Number analyzed (Participants) | 142
percentage change
  Mean change in CTX from baseline to month 3 | 49 (43)
  Mean change in CTX from baseline to month 6 | 64 (62)
  Mean change in TH BMD from baseline to month 12 | 1.14 (0.14)

2. Secondary Outcome: Percent Change in Bone Turnover Markers Measured Three and Six Months After Stopping Alendronate Treatment and BMD After One and Two Years
Description: We constructed receiver operating characteristic (ROC) curves to evaluate if changes in p-CTX or p-PINP measured three and six months after stopping alendronate predicted TH BMD loss above the least significant change at month 12 and/or month 24 at the individual level.
Time Frame: one and two years after baseline
Population: None of the ROC curves investigating the ability of change in bone turnover markers to predict BMD loss beyond LSC at any site at month 12 or month 24 at the individual level had AUC above 60% meaning that it was not possible to identify a specific cut-off value that could predict significant bone loss at the individual level.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Study Population
Number analyzed (Participants) | 142
percentage change
  Mean change in PINP from baseline to month 3 | 36 (40)
  Mean change in PINP from baseline to month 6 | 54 (45)
  Mean change in TH BMD from baseline to month 12 | -1.14 (0.14)
  Mean change in TH BMD from baseline to month 24 | -2.65 (0.39)

3. Secondary Outcome: Number of Participants in Which CTX Increased Above the Least Significant Change
Description: Number of participants in which CTX increased above the least significant change.
  The Department of Clinical Biochemistry, Rigshospitalet, Glostrup, Denmark provided the the least significant change for p-CTX > 30%.
Time Frame: From baseline to month 24
Measure: Number; unit: participants
Arm/Group | Study Population
Number analyzed (Participants) | 124
participants | 85

4. Secondary Outcome: The Number of Participants Who Lost BMD Beyond the Least Significant Change (LSC) at the Lumbar Spine and Total Hip.
Description: the number of patients who lost BMD beyond the LSC at the lumbar spine (>3%) and total hip (>5%)
Time Frame: from baseline to month 24
Measure: Number; unit: participants
Arm/Group | Study Population
Number analyzed (Participants) | 124
participants
  Spine | 21
  Total hip | 26

5. Secondary Outcome: If Baseline Bone Turnover Markers at the Time of Alendronate Discontinuation Predict Changes in BMD After One and Two Years.
Description: We constructed receiver operating characteristic (ROC) curves to evaluate if baseline p-CTX or baseline p-PINP at the time of alendronate discontinuation predicted TH BMD loss above the least significant change at month 12 and/or month 24 at the individual level.
Time Frame: Changes in TH BMD after one and two years.
Population: None of the ROC curves investigating the ability of baseline bone turnover markers to predict BMD loss beyond LSC at any site at month 12 or month 24 at the individual level had AUC above 60% meaning that it was not possible to identify a specific cut-off value that could predict significant bone loss at the individual level.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Study Population
Number analyzed (Participants) | 142
percentage change
  Mean change in TH BMD after one year | -1.14 (0.14)
  Mean change in TH BMD after two years | -2.65 (0.39)

ADVERSE EVENTS:
Time Frame: From baseline to month 24
Groups:
- Study Population: Postmenopausal women (postmenopausal for at least 2 years) and men above 50 years, who had been treated with ALN for at least five years and had a THBMD T-score > -2.5 and LSBMD (L1-L4) T-score > -4.
  We excluded patients with any low-energy fracture within the previous 5 years during ALN treatment (not including fingers, toes, or skull), low-energy VFx or hip fracture at any time, on-going treatment with systemic glucocorticoids, metabolic bone disease, hormone replacement therapy, cancer and other conditions affecting bone metabolism.
Arm/Group | Study Population
All-Cause Mortality (participants affected / at risk) | 0/142
Serious Adverse Events (participants affected / at risk) | 7/142
Other Adverse Events (participants affected / at risk) | 68/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Population (N=142)
Cancer (Investigations) | 7 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Population (N=142)
Fracture (Musculoskeletal and connective tissue disorders) | 15 (15)
Arrhythmia, acute myocardial infarction, hypertension (Cardiac disorders) | 10 (10)
Cataract, glaucoma (Eye disorders) | 9 (9)
Lower urinary symptoms, infection and kidney stones (Renal and urinary disorders) | 9 (9)
Arthralgia, osteoarthritis, back pain (Musculoskeletal and connective tissue disorders) | 15 (15)
Upper and lower respiratory tract infection, pneumonia, bronchitis (Respiratory, thoracic and mediastinal disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT03051620/Prot_SAP_000.pdf